CLINICAL TRIAL: NCT03176940
Title: 2-Hydroxybenzylamine: Initial Evaluation in Humans
Brief Title: 2-HOBA: Initial Evaluation in Humans
Acronym: 2-HOBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metabolic Technologies Inc. (Industry)
Collaborators: Vanderbilt University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, John Rathmacher, PhD, Director of Clinical Research, Metabolic Technologies Inc.
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 161861; R44AG055184 (NIH)
Record Dates: First submitted 2017-04-20; First posted 2017-06-06 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Healthy Volunteers
Keywords: Escalating Dosage
MeSH Terms: interventions — 2-(aminomethyl)phenol

STUDY DESIGN:
Intervention Model Description: The 3+3 design will be employed for this trial. At least 3 volunteers will be studied at each dose level and evaluated for adverse effects. If 0 of 3 volunteers experiences adverse events (AE), the dose is escalated. If 1 of 3 volunteers experiences an AE, 3 additional volunteers are treated. If none of the additional volunteers develop an AE, the dose is escalated, otherwise escalation ceases. If 2 of 3 or 2 of 6 volunteers experience an AE, the maximum tolerated dose (MTD) has been exceeded.
Who Masked: Participant, Care Provider
Masking Description: The dietary supplement will be delivered to the Clinical Research Center by the Investigational Pharmacy at Vanderbilt University Medical Center. Staff nurses and participants will be blinded to the capsule dosage content.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 2-HOBA first dose (Experimental): Dose escalation studies in humans: 50mg dose
  Interventions: Dietary Supplement: 2-HOBA
- 2-HOBA second dose (Experimental): Dose escalation studies in humans: 100mg dose
  Interventions: Dietary Supplement: 2-HOBA
- 2-HOBA third dose (Experimental): Dose escalation studies in humans: 200mg dose
  Interventions: Dietary Supplement: 2-HOBA
- 2-HOBA fourth dose (Experimental): Dose escalation studies in humans: 330mg dose
  Interventions: Dietary Supplement: 2-HOBA
- 2-HOBA fifth dose (Experimental): Dose escalation studies in humans: 550mg dose
  Interventions: Dietary Supplement: 2-HOBA
- 2-HOBA sixth dose (Experimental): Dose escalation studies in humans: 825mg dose
  Interventions: Dietary Supplement: 2-HOBA

INTERVENTIONS:
Dietary Supplement: 2-HOBA — 2-HOBA is a compound found in buckwheat and is given as 2-HOBA acetate
  Other Names: 2-Hydroxylbenzylamine

SUMMARY:
The purpose of this study is to evaluate the administration of single doses of 2-HOBA in humans, with an escalation of doses that begins with the calculated Maximum Recommended Starting Dose. This evaluation will assess tolerability to oral administration of 2-HOBA, obtain pharmacokinetic data, characterize the 2-HOBA metabolic pathways, and determine the relation of dose to prevention of formation of bi-functional electrophile adducts in blood. Characterization of the metabolic fate of 2-HOBA will be supported by investigations that evaluate metabolism in microsomes and cells.

DETAILED DESCRIPTION:
Consenting volunteers of at least 18 years old with no morbidity, including males, and females who are not pregnant will be recruited for the study. A maximum of 28 volunteers may be enrolled with a reasonable sampling of ethnicities from the Nashville area, and an effort will be made to recruit equal numbers of males and females. Additionally, an effort will be made to study as old a population as possible and to recruit relatively similar age groups for males and females. All volunteers will be admitted to the Vanderbilt Clinical Research Center (CRC) as inpatients.

A complete health history and physical examination will be conducted by a physician. Volunteers will be asked to collect and bring their first morning voided urine for baseline urinalysis. An EKG, baseline blood analysis, vital signs, and questions about feelings and adverse events will be asked prior to supplement administration. All tests will be repeated at various intervals throughout the 24-hour study period. A physician will oversee all clinical aspects of the study and will be responsible for all trial-related medical decisions. Pharmacokinetics will be studied through the blood analyses at intervals throughout the study and 24-hour urine collection after administration of the supplement.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals older than 18;
* Males and females who are not pregnant at the time of the study; and
* Not taking any medication 2 weeks prior to and during the study.

Exclusion Criteria:

* Inability to give informed consent;
* Diseases that could manifest symptoms or signs that would confound interpretation of the relation between drug action and potential adverse effects;
* Diseases that could manifest morbidity;
* Known cardiac disease, kidney disease, or hepatic dysfunction;
* The need to discontinue any drug that is administered as standard of care treatment; and
* Unwillingness or inability to use approved birth-control methods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Dose Tolerability | 24 hours
  Tolerability will be assessed by occurrence of Adverse Events (AEs). If AEs occur in 2 out of 6 volunteers, the dose will be declared not tolerated and the previous dose with no AEs will be declared maximum tolerable dose.
  AEs < 2: dose is tolerated AEs ≥ 2: dose is not tolerated

CONTACTS AND LOCATIONS:
Overall Officials: John A Rathmacher, PhD, Principal Investigator — Metabolic Technologies Inc.
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pitchford LM, Rathmacher JA, Fuller JC Jr, Daniels JS, Morrison RD, Akers WS, Abumrad NN, Amarnath V, Currey PM, Roberts LJ, Oates JA, Boutaud O. First-in-human study assessing safety, tolerability, and pharmacokinetics of 2-hydroxybenzylamine acetate, a selective dicarbonyl electrophile scavenger, in healthy volunteers. BMC Pharmacol Toxicol. 2019 Jan 5;20(1):1. doi: 10.1186/s40360-018-0281-7. PMID 30611293